CLINICAL TRIAL: NCT05027945
Title: A Phase II Study of Allogeneic Hematopoietic Stem Cell Transplant for Subjects With VEXAS (Vacuoles, E1 Enzyme, X-linked, Autoinflammatory, Somatic) Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000404; 000404-C
Record Dates: First submitted 2021-08-28; First posted 2021-08-31 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11-24

CONDITIONS: Immunodeficiency; Hematopoietic Stem Cell Transplantation
Keywords: Immune Dysregulation; Haploidentical; hematoinflammatory diseases; Myelodysplastic Syndromes; Autoimmune Disorders
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Myelodysplastic Syndromes; Autoimmune Diseases | interventions — Mycophenolic Acid; Tacrolimus; Busulfan; Whole-Body Irradiation; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm A (Experimental): Reduced intensity regimen (Fludarabine, busulfan)+HSCT+GVHD prophylaxis
  Interventions: Procedure: Allogeneic HSCT; Drug: Busulfan test dose; Drug: Mycophenolate mofetil (MMF); Drug: Tacrolimus; Drug: Busulfan; Drug: Fludarabine; Drug: Post-Transplant Cyclophosphamide (PTCY)
- Arm B (Experimental): Reduced intensity regimen (Fludarabine, low dose cyclophosphamide, 200cGY TBI, busulfan)+HSCT+GVHD prophylaxis
  Interventions: Procedure: Allogeneic HSCT; Drug: Busulfan test dose; Drug: Mycophenolate mofetil (MMF); Drug: Tacrolimus; Drug: Busulfan; Radiation: Total Body Irradiation (TBI); Drug: Fludarabine; Drug: Cyclophosphamide (CY); Drug: Post-Transplant Cyclophosphamide (PTCY)

INTERVENTIONS:
Procedure: Allogeneic HSCT — stem cell transplant on day 0
Drug: Busulfan test dose — 0.8 mg/kg IV over 2 hours. May be skipped if real-time PKs are done during conditioning.
Drug: Mycophenolate mofetil (MMF) — Mycophenolate mofetil (MMF): 15 mg/kg IV over 2 hours BID starting on day +5 until approximately day +35 (+/-2 days)
Drug: Tacrolimus — Starting on day +5, start at 0.02 mg/kg IV continuous infusion over 24 hours until day +180 and titrated to trough levels of 5-15 mg/ml.
Drug: Busulfan — AUC Targeted Dose based on busulfan test dose PKs, IV infusion over 3 hours once daily (3.2 mg/kg IV per day will be the default dose) per the below time frame: For 8/8 Matched Related or Unrelated Donor Busulfan dose will be on days -6, -5, and -4 For 7/8 Matched Related or Unrelated or Haploidentical Donor Busulfan dose will be on days -4 and -3
Radiation: Total Body Irradiation (TBI) — For 7/8 Matched Related or Unrelated or Haploidentical Donor, 200cGy on day -1
  Arms: Arm B
Drug: Fludarabine — 40 mg/m2 IV over 30 mins daily For 8/8 Matched Related or Unrelated Donor Fludarabine dose will be on days -6, -5, -4, and -3 For 7/8 Matched Related or Unrelated or Haploidentical Donor Fludarabine dose will be on days -6, -5, -4, -3, and -2
Drug: Cyclophosphamide (CY) — For 7/8 Matched Related or Unrelated or Haploidentical Donor, prior to transplant 14.5 mg/kg IV daily on days -6 and -5
  Arms: Arm B
Drug: Post-Transplant Cyclophosphamide (PTCY) — Post-Transplant Cyclophosphamide: 50 mg/kg IV daily over 2 hours on days +3 and +4, dosed according to ideal body weight

SUMMARY:
Background:

Allogeneic hematopoietic stem cell transplant involves taking blood stem cells from a donor and giving them to a recipient. The transplants are used to treat certain diseases and cancers. Researchers want to see if the transplant can treat VEXAS Syndrome.

Objective:

To see if stem cell transplants can be successfully performed in people with VEXAS and even improve the disease.

Eligibility:

People ages 18-75 who have VEXAS Syndrome that has caused significant health problems and standard treatment either has not worked or is not available.

Design:

Participants will be screened with:

Physical exam

Medical review

Blood and urine tests

Heart and lung function tests

Bone marrow biopsy

Participants will have a chest x-ray. They will have an imaging scan of the head, chest, abdomen, pelvis, and sinus. They will have a bone density scan. They will have a dental exam and eye exam. They will meet with specialists. They will repeat some screening tests.

Participants will be admitted to the NIH hospital. They have a central venous catheter put into a vein in the chest or neck. They will receive drugs to prepare their bone marrow for the transplant. They may have total body irradiation. They will receive the donor stem cells through the catheter. They will get other drugs to prevent complications and infections. After discharge, they must stay in the DC area for 3 months for weekly study visits.

Participants will have study visits 30, 60, 100, 180, 210, 240, 300, and 360 days later. After that, they will have yearly visits for 2 years and then be contacted yearly by phone....

DETAILED DESCRIPTION:
Background:

* In 2019, investigators at the National Institutes of Health defined a new disease syndrome named VEXAS: Vacuoles in bone marrow cells, E1 enzyme mutations, X-linked, Autoinflammatory, Somatic syndrome. This syndrome is characterized by inflammatory and hematologic features and is frequently accompanied by marrow dysplasia, progressive bone marrow failure, and in some cases, the development of overt myelodysplastic syndrome (MDS) or other myeloid neoplasms. Somatic mutations are present at methionine 41 in UBA1, an X-linked gene encoding the major E1 ubiquitin activating enzyme that initiates the majority of cellular ubiquitylation.
* The inflammatory features of VEXAS include fever, pulmonary infiltrates, skin lesions, ear and nose chondritis, musculoskeletal involvement, and elevated inflammatory markers. The hematologic features include cytopenia, characteristic vacuoles in myeloid and erythroid precursors cells, and dysplastic bone marrow. Patients included in the initial description of the syndrome fulfill clinical or classification criteria for both inflammatory diseases (relapsing polychondritis, Sweet syndrome, polyarteritis nodosa, giant cell arteritis) and hematologic conditions (MDS, myeloid neoplasms or plasma cell dyscrasia). The inflammatory features of VEXAS are refractory to treatment other than high doses of glucocorticoids. Increased mortality and frequent morbidity are common in VEXAS secondary to the disease and treatment-related complications. The clinical manifestations of VEXAS are time-dependent. Systemic inflammation typically precedes progressive bone marrow failure with or without the development of hematologic malignancies leading to death. Escalating doses of glucocorticoids are typically administered to control the refractory, progressive features of systemic inflammation. Worsening cytopenias often require transfusion support.
* The discovery of hematologic mosaicism as the genetic driver of rheumatologic/hematologic syndromes defines a novel class of diseases, termed hematoinflammatory diseases (HINDS), and it raises the possibility that therapies aimed at eradicating these clones may be efficacious in this patient population.

Objectives:

Primary Objectives:

* To determine whether allogeneic hematopoietic stem cell transplantation (HSCT) results in sustained donor engraftment at day 100 and one-year post-HSCT.
* To determine whether allogeneic HSCT results in reversal of the clinical phenotype of VEXAS at one year and two years post-HSCT without requiring interval prednisone at >= 0.5 mg/kg per day for reasons other than graft-versus-host disease (GVHD).

Eligibility:

* Recipients ages 18-75 year-old with or without a somatic mutation in UBA1 who have: 1) the clinical phenotype for VEXAS with refractory cutaneous, pulmonary, musculoskeletal, and/or other recurrent acute inflammatory manifestations, and 2) require >= 0.5 mg/kg per day of prednisone for inflammatory manifestations OR have cytopenia (transfusion dependent anemia, transfusion dependent thrombocytopenia/platelets <75,000, neutropenia <1,000/microL) or myeloid neoplasm (by WHO criteria) or being intolerant or refractory to use steroids.
* Have an 8/8 or 7/8 HLA-matched related or unrelated donor, or a haploidentical related donor.

Design:

-For Recipients with 8/8 HLA Matched Donors:

Participants will receive reduced intensity conditioning with the following regimen:

fludarabine 40 mg/m^2 IV once daily for four days on days -6, -5, -4, -3 and Busulfan IV for three days on days -6, -5, -and -4 followed by HSCT on day 0. The busulfan dose will be based on pharmacokinetic levels from the test dose and/or real time PKs and will be targeted to AUC of 2500-3500 microMol*min/L (31-43 mg*h/L) (2.5 - 2.8 mg/kg IV may be used on D-6 with real time PK for D-5 and D-4).

-For Recipients with 7/8 HLA Matched Donors or Haploidentical Related Donors:

Participants will receive reduced intensity conditioning with the following regimen:

fludarabine 30 mg/m^2 IV once daily for five days on days -6, -5, -4, -3, and -2, cyclophosphamide 14.5 mg/kg for two days on days -6 and -5, 200 cGy total body irradiation (TBI) on day -1, busulfan IV once daily for two days on days -4 and -3, and HSCT on day 0. The busulfan dose will be based on pharmacokinetic levels from the test dose and/or real time PKs and will be targeted to an AUC of 2500-3500 microMol*min/L (21-29 mg*h/L) (2.5 -2.8 mg/kg IV per day may be used on D-4 with real time PK for D-3).

-For Post-Transplant GVHD Prophylaxis:

Post-transplant GVHD prophylaxis in all groups will consist of cyclophosphamide 50 mg/kg IV once daily for 2 days on days +3 and +4, along with mycophenolate mofetil from day +5 to approximately day +45 and tacrolimus from day +5 to approximately day +180.

ELIGIBILITY:
* INCLUSION CRITERIA:

Non-disease related

* Age >= 18-year-old and <= 75-year-old
* Availability of an 8/8 or 7/8 HLA-matched related or unrelated donor, or a haploidentical related donor
* Karnofsky performance status of >= 40%
* Adequate end-organ function, defined as follow:

  1. Left ventricular ejection fraction > 35%, preferably by 2-D echocardiogram (ECHO) obtained within 60 days prior to treatment initiation.
  2. Creatinine <= 2.0 mg/dl and creatinine clearance >= 30 ml/min;
  3. Serum conjugated bilirubin < 3.0 mg/dl; serum ALT and AST <= 5 times upper limit of normal.
* Pulmonary function tests: FEV1 and DLCO >30%
* Ability of subject to understand and the willingness to sign a written informed consent document.
* As therapeutic agents used in this trial may be harmful to a fetus, individuals of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at the study entry and for at least one-year post-allo HCT. Should an individual become pregnant or suspect they are pregnant while she or her partner is participating in the study, she should inform her treating physician immediately.
* Willingness to remain in the NIH hospital or, if discharged, live within 2 hours drive from the NIH, for a minimum of 100 days after transplant or longer, if there are complications. If outpatient in the first 100 days after transplant, participant must commit to having an adult caregiver with them at all times.

Disease related

* Somatic mutation in UBA1 performed by a CLIA or CAP certified laboratory. NOTE: Participants without a mutation or unknown mutation status may be eligible if they have a clinical history that is characteristic of an individual with VEXAS syndrome including two or more of a-e below.
* Inflammatory clinical phenotype for VEXAS syndrome with at least one VEXAS disease manifestation below:

  1. constitutional symptoms including fevers, fatigue, and weight loss
  2. cutaneous symptoms of VEXAS including biopsy proven neutrophilic dermatosis, cutaneous vasculitis, periorbital inflammation
  3. pulmonary symptoms of VEXAS with pulmonary infiltrates, pleural effusion
  4. musculoskeletal or cartilaginous involvement including inflammatory arthritis, ear chondritis, and nasal chondritis
  5. inflammatory disease in other major organ systems including cardiac, gastrointestinal, ocular, etc.
* Presence of cytopenia defined as at least one of the following:

  i. Absolute neutrophil count <=1000/ microliter

ii. platelet count <= 75,000/microliter or platelet transfusion dependence (at least 4 platelet transfusions in the 8 weeks prior to study entry

iii. hemoglobin <= 10.0g/dL or red cell transfusion-dependence (at least 4 units of PRBCs in the 8 weeks prior to treatment initiation) or meeting criteria for myeloid neoplasm (MN) by updated 2022 WHO criteria or 2022 International Consensus Classification (ICC) of myeloid neoplasms and acute leukemia

OR:

-Participants who have failed standard medical management (requiring >= 0.5mg/kg per day of prednisone for the above listed inflammatory condition or intolerance or refractory to use of corticosteroids and/or steroid sparing medications as well as biological response modifiers over the last 6 months), or when no standard medical treatment is available.

EXCLUSION CRITERIA:

* HCT Comorbidity Index >= 5. Note: Comorbidities that are specifically addressed in the inclusion criteria will not be included in the calculation of HCT-CI score.
* Participants with multiple myeloma. Note: participants with low risk smoldering multiple myeloma or monoclonal gammopathy of unknown significance will not be excluded)
* Participants who are receiving any other investigational agents within the last 30 days before treatment initiation.
* HIV-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents (steroids, cyclophosphamide, busulfan, tacrolimus, MMF, filgrastim or filgrastim biosimilar) used in the study.
* Pregnant individuals are excluded from this study because the study agents have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study agents, breastfeeding should be discontinued if the mother is treated with the study agents.
* Uncontrolled intercurrent illness or social situations (as determined by a licensed master social worker) that would limit compliance with study requirements.
* Presence of active uncontrolled infections that in the opinion of the PI would make it unsafe to proceed with transplantation.
* Active psychiatric disorder which is deemed by the PI to have significant risk of compromising compliance with the transplant protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Reversal of clinical phenotype of VEXAS | +1 and +2 years post HSCT
  fraction of subjects who achieve complete clinical response without use of additional glucocorticoid therapy and without steroid-sparing therapy
Sustained donor engraftment | day +100 and +1 year post HSCT
  defined as neutrophil recovery with ANC = 500/mm^3 for 3 consecutive days associated with > 50% T-cell and myeloid cell donor chimerism at day 100 and one year post-HSCT

SECONDARY OUTCOMES:
Safety of allo HSCT | +1, +2 and +3 years post HSCT
  Transplant-related toxicity will include if allogeneic HSCT in participants with VEXAS results in the absence of secondary graft failure. The fraction of participants who have secondary graft failure will be reported along with a 95% two-sided confidence interval, separately by cohort.
incidence of grade III-IV acute GVHD and moderate to severe chronic GVHD | +1 and +2 years post HSCT
  group comparison of participants with an 8/8 HLA matched related or unrelated donor compared to group of participants with 7/8 HLA matched related or unrelated donor or haploidentical donor. Reported with 95% two-sided confidence intervals. The fractions will also be reported separately by cohort using simple estimates along with 95% two-sided confidence intervals. In addition cumulative incidence curves along with a 95% two-sided confidence interval.
Overall survival and event free survival | +1, +2 and +3 years post HSCT
  Overall and event free survival will be determined using Using the Kaplan-Meier method, along with the median value and the 95% confidence interval at the median, separately by cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Ajoy L Dias, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGAP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- [Derived] Fiumara M, Campochiaro C, Molteni R. Decoding VEXAS syndrome: emerging insights into pathogenesis and clinical management. Curr Opin Rheumatol. 2026 Jan 1;38(1):45-52. doi: 10.1097/BOR.0000000000001137. Epub 2025 Nov 5. PMID 41175032
- [Derived] Koster MJ, Samec MJ, Warrington KJ. VEXAS Syndrome-A Review of Pathophysiology, Presentation, and Prognosis. J Clin Rheumatol. 2023 Sep 1;29(6):298-306. doi: 10.1097/RHU.0000000000001905. Epub 2022 Oct 17. PMID 36251488
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000404-C.html